CLINICAL TRIAL: NCT06987240
Title: Comparison Of Ultrasound-Assisted Combined Spinal Epidural Procedure With Anatomical Landmark Method In Obese Patients Undergoing Lower Extremity Surgery
Brief Title: Landmark vs Ultrasound For Combined Spinal Epidural
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-SEAH-BC-KSEA
Record Dates: First submitted 2025-04-22; First posted 2025-05-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Obesity (Body Mass Index >30 kg/m2); Ultrasonography; Combined Spinal Epidural Anesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasonography (USG) (Active Comparator): In this group, patients will first be marked with ultrasonography and the time required for this procedure will be recorded. Then, the needle will be inserted from the marked area. When performing the combined spinal epidural procedure, the number of needle insertions, the number of directions will be recorded and the time from needle insertion to needle exit will be recorded.
  Interventions: Procedure: Ultrasonography-guided combined spinal epidural anesthesia application
- Landmark (L) (Placebo Comparator): Patients in this group will be marked according to anatomical landmarks. The time from needle entry to exit and the number of needle entries and directions will be recorded.
  Interventions: Procedure: Combined spinal epidural anesthesia with Landmark

INTERVENTIONS:
Procedure: Ultrasonography-guided combined spinal epidural anesthesia application — patients with BMI>30
  Arms: ultrasonography (USG)
Procedure: Combined spinal epidural anesthesia with Landmark — Patients with BMI>30
  Arms: Landmark (L)

SUMMARY:
A comparison of two different methods used in routine anesthesia practices will be made for the insertion of a catheter that will be placed at the waist for anesthesia in obese patients who will undergo orthopedic surgery.

60 obese patients aged 40-80, ASA II-III, BMI>30, who are planned to undergo elective orthopedic lower extremity surgery by placing a combined spinal epidural catheter at Sakarya University Medical Faculty Education and Research Hospital will be included in the study.

General anesthesia or regional anesthesia techniques are routinely used in lower extremity surgery in our clinic. When placing a combined spinal epidural catheter, the entry site is determined by looking at anatomical landmarks or using ultrasound.

Patients will be divided into two different groups as Anatomical Marking or Ultrasound.

Patients in the Ultrasound group will be taken to the block room in our operating room before the operation and a location marking will be performed with Ultrasound in the block room.

Patients in the Anatomical Marking group will be brought to a sitting position in the operating room in the operating room and a location marking will be performed by hand examination.

After determining the needle entry site, patients in both groups will undergo the Combined spinal epidural catheter placement procedure, which is performed routinely under sterile conditions, and the success rate at the first attempt, total success rates, number of needle redirections, and complications during the procedure will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III
* BMI>30
* Elective orthopedic lower extremity surgery
* Combined spinal epidural anesthesia (CSEA)

Exclusion Criteria:

* Patients with CSEA contraindication
* ASA IV-V
* Diagnosed with scoliosis
* Patients with anatomical disorders
* Patients who did not agree to participate in the study
* Patients for whom follow-up conditions could not be met

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | up to 20 weeks
  FIRST TRY SUCCESS; will be defined as FINDING THE EPIDURAL SPACING WITHOUT REMOVING THE NEEDLE FROM THE SKIN.

SECONDARY OUTCOMES:
Number of needle insertions | up to 20 weeks
  Number of referrals after needle intervention
Time to determine the needle insert | up to 20 weeks
  Duration of determination of the needle insertion site by ultrasonography or anatomical landmarks
Total procedure time | up to 20 weeks
  Procedure time: The time from the entry of the Tuohy needle through the skin to the completion of the procedure, placement of the catheter and withdrawal of the needle

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University Hospital, Sakarya, Adapazarı, Turkey (Türkiye)